CLINICAL TRIAL: NCT00004378
Title: Stem Cell Transplantation (SCT) for Genetic Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, Los Angeles (Other)
Purpose: Treatment
Other Study IDs: 199/11981; UCLA-92010034
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2002-04

CONDITIONS: Thrombocytopenia; Metachromatic Leukodystrophy; Fanconi's Anemia; Thalassemia Major; Pure Red-Cell Aplasia; Inborn Errors of Metabolism
Keywords: Fanconi's anemia; amegakaryocytic thrombocytopenia; aplastic anemia; congenital pure red cell aplasia; genetic diseases and dysmorphic syndromes; hematologic disorders; inborn errors of metabolism; metachromatic leukodystrophy; pure red cell aplasia; rare disease; sphingolipidoses; thalassemia major
MeSH Terms: conditions — Thrombocytopenia; Leukodystrophy, Metachromatic; Fanconi Anemia; beta-Thalassemia; Red-Cell Aplasia, Pure; Metabolism, Inborn Errors; Anemia, Aplastic; Anemia, Diamond-Blackfan; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases; Sphingolipidoses | interventions — Stem Cell Transplantation

INTERVENTIONS:
Procedure: Stem Cell Transplantation

SUMMARY:
OBJECTIVES: I. Ascertain whether stem cell transplantation (SCT) is an effective method by which missing or dysfunctional enzymes can be replaced in patients with various inborn errors of metabolism.

II. Determine whether clinical manifestations of the specific disease may be arrested or reversed by this treatment.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive either cyclophosphamide and high dose total body irradiation (TBI) or busulfan and cyclophosphamide.

Cyclophosphamide IV is given on days -5 and -4 and TBI on days -2, -1, and 0. Busulfan is given orally every 6 hours on days -9 through -6 and cyclophosphamide IV on days -5 through -2. Patients rest on day -1.

Patients receive bone marrow infusion on day 0. For GVHD prophylaxis, patients receive methotrexate on day 1, then on days 3, 6, and 11. Cyclosporine IV begins on day -2 over 12 hours, followed by continuous infusion for 21 days. Then, oral doses of cyclosporine are given every 12 hours to patients who tolerate oral feeding. Cyclosporine is continued 6 months posttransplant, then tapered 10% per week and stopped.

Patients who receive genotypically HLA nonidentical stem cells undergo additional GVHD prophylaxis with methylprednisolone (IV or PO) or its equivalent every 12 hours on days 3 to day 100. Dose is then tapered as tolerated over 1 month.

Patients who receive cord blood stem cells receive methylprednisolone instead of methotrexate for GHVD prophylaxis. Methylprednisolone is given 3 times daily beginning on day 5 and continuing until day 17. Then, methylprednisolone is tapered 10% per week as clinically tolerated.

To accelerate engraftment, patients receive filgrastim IM daily beginning on day +1 and continuing until ANC equals 5000.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Hereditary enzymopathies, such as: Metachromatic leukodystrophy
* Congenital Immunodeficiencies
* Heritable hematologic disorders, such as: Thalassemia major Refractory Diamond-Blackfan anemia Fanconi anemia Amegakaryocytic thrombocytopenia

--Patient Characteristics--

* Age: Under 18
* Other: SCT is performed using a histocompatible related donor, an unrelated donor, or an unrelated cord blood donor Haploidentical donors are accepted for patients with severe congenital immunodeficiency

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Stephen A. Feig, Study Chair — University of California, Los Angeles
Locations (1):
- University of California Los Angeles Medical Center, Los Angeles, California, United States